CLINICAL TRIAL: NCT06317090
Title: Vertical Guided Bone Regeneration: LPRF Block vs a Mixture of Autogenous Bone With Deproteinized Bovine Bone Mineral. A Split-mouth RCT Study With 25 Months Follow-up
Brief Title: Vertical GBR LPRF Block vs. Autogenous Bone With DBBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Ana CASTRO SARDA, prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S59813-2
Record Dates: First submitted 2023-06-06; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Bone Resorption

STUDY DESIGN:
Intervention Model Description: split-mouth 2 arm RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: neither the patient, nor the outcome assessor was aware at which side which grafting material was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): LPRF block as a grafting material
  Interventions: Procedure: guided bone regeneration
- Control (Experimental): 50% autogenous bone, 50% DBBM as a grafting material
  Interventions: Procedure: guided bone regeneration

INTERVENTIONS:
Procedure: guided bone regeneration — a non-resorbable membrane was used as a space maintainer, filled with a particulated bone graft.
  Other Names: GBR

SUMMARY:
split-mouth RCT, 25 months follow up. GBR protocol with LPRF as grafting material in the test group and autogenous bone with DBBM as grafting material in the control group.

DETAILED DESCRIPTION:
6 patients were included in this split-mouth RCT. In control sites a horizontal GBR procedure was performed using a titanium reinforced dPTFE membrane with a graft consisting of 50% autogenous bone and 50% DBBM. In test sites a titanium reinforced dPTFE membrane was used, with a graft consisting of an LPRF block. This was left to heal for 9 months. Subsequently an implant was placed. At time of implant placement a bone biopsy was taken. After 4 months of osseointegration the abutment connection was performed. 1 year after loading of the implants a final check was done. CBCT scans were taken at intake, immediately after reconstruction, 9 months after reconstruction, before implant placement and 1 year after loading of the implants.

Primary outcome measure is the bone volume as measured on the CBCT scans. Secondary outcome measures are bone quality in the biopsy, buccal bone thickness around the oral implant, number and type of complications, cumulative survival rates of the implants 1 year after loading.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, with ASA I or II, between 18 and 80 years old
* 2 implant sites requiring vertical bone augmentation prior to implant placement
* Both sites in the same jaw
* Good general health as documented by self-assessment

Exclusion Criteria:

* Any systemic medical condition that could interfere with the surgical procedure, planned treatment or healing of the patient
* Immunosuppression, Diabetes, Anticoagulation or Antiaggregatory medication.
* Current pregnancy or breast feeding/ lactating at the time of recruitment.
* Radiotherapy or Chemotherapy in head and neck area.
* Intravenous and oral bisphosphonate therapy.
* Smoking
* Unwillingness to return for the follow-up examination.
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unrealistic expectations
* Presence of osseous pathologies, that might interfere with normal wound healing
* Presence of oral lesions (such as ulceration, malignancy)
* Local inflammation, including untreated periodontitis
* Patients with inadequate oral hygiene or unmotivated for adequate home care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
bone volume as measured on CBCT scans | CBCT scans at intake, with follow-up until 25 months post-operative
  CBCT scans taken and software used for measurement

SECONDARY OUTCOMES:
Buccal bone thickness around the implants | CBCT scans at placement of the implant and 1 year after loading of the implant
  Bone thickness measured on CBCT scans
Buccal bone thickness around the implants | CBCT scans at 1 year after loading of the implant
  Bone thickness measured on CBCT scans
Cumulative survival rate of the implants | 16 months of follow-up
  Implants followed for 1 year after loading and survival recorded
rates and types of complications | 25 months
  All complications recorded during 25 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
all info available on request